CLINICAL TRIAL: NCT02152878
Title: Transcranial Direct Current Stimulation for the Treatment of Bipolar Depression
Acronym: TDCS-BD
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Brain & Behavior Research Foundation (Other)
Responsible Party: Principal Investigator, Andre Brunoni, MD, PhD, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BETTER
Record Dates: First submitted 2014-05-29; First posted 2014-06-02 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Depression, Bipolar
Keywords: transcranial direct current stimulation; non invasive brain stimulation; bipolar disorder; depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active stimulation (Active Comparator): Active stimulation (tDCS) will be used in the dose of 2mA /30 min per day, for 10 days and two extra sessions every other week (total of 12 sessions).
  Interventions: Device: Active stimulation
- Sham stimulation (Placebo Comparator): For Sham Transcranial Direct Current Stimulation, the device is automatically turned off after 30 seconds of stimulation and remains turned off.
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Sham stimulation — For sham tDCS, the device will be turned off after 30 seconds of stimulation.
  Other Names: TDCS
  Arms: Sham stimulation
Device: Active stimulation — For active tDCS, we will place the anode and the cathode over the left and right dorsolateral prefrontal cortex areas, respectively (corresponding to F3 and F4 according to the EEG 10-20 system). We will use 5x5 cm electrodes and a 2mA current for 30 minutes per day. This montage is known as "bifrontal" setup and has been previously used in major depression trials
  Arms: Active stimulation

SUMMARY:
Non-invasive brain stimulation therapies have been increasingly investigated in recent years as a treatment for neuropsychiatric disorders, particularly mood disorders. They are particularly appealing since many patients are either refractory or present side effects to standard pharmacological regimens. TDCS (transcranial direct current stimulation). a novel non- pharmacological brain stimulation technique, might help in overcoming some of these issues, since it has low cost, high portability and it is relatively easy to use. TDCS consists in applying a weak, direct current through two electrodes placed over the scalp; the anode and the cathode increasing and decreasing cortical excitability during and beyond the period of stimulation. It is also a safe technique with only mild adverse effects described. Previous studies, some of them from our group, have described that tDCS is an effective technique for major depression. However, the role of tDCS as a treatment for bipolar depression (BD) has been insufficiently investigated. Therefore, our aim is to address the antidepressant effects of tDCS in BD in a randomized, sham- controlled trial in a refractory sample.

DETAILED DESCRIPTION:
BD represents the greatest burden on patients with bipolar disorder, since the depressive episodes are the most frequent and also particularly associated with suicide 7. BD treatment is controversial, with some stricter guidelines recommending only lithium, lamotrigine and quetiapine as a first-treatment, whereas others allow the use of antidepressants (which can increase manic switch and should be used in association with mood stabilizers) and other anticonvulsants and antipsychotics 8. For refractory BD the available level I evidence is very scarce, with only seven studies exploring this issue hitherto 9. Therefore, the importance of this study proposal is justified considering the burden of the disease, the paucity of current therapeutic studies and the promising results presented for tDCS in unipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* bipolar depressed (type I, II or not otherwise specified) participants with symptoms in spite of an adequate treatment course with mood stabilizers.
* the depressive episode has to be of at least moderate intensity (baseline HDRS>=16)
* read and understand Portuguese

Exclusion Criteria:

* other neuropsychiatric conditions, such as schizophrenia, substance dependence, dementias, traumatic brain injury, epilepsy and so forth (although participants with anxiety disorders can be included whether the primary diagnosis is BDD);
* mixed states, defined as simultaneously presenting (hypo)manic symptoms with a Young Manic Rating Scale (YMRS) > 8;
* pregnancy;
* specific contra-indications to tDCS;
* severe/life-threatening clinical conditions. Participants will have to be drug-free or at stable drug regimen for at least 6 weeks prior to trial onset. Benzodiazepine drugs will be allowed, although only at low doses (less than 20mg/day of diazepam or equivalent).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Change in Hamilton Scale for Depression, 17 items | week 0 (baseline), week 2, week 4 and week 6 (endpoint)
  Continuous measure (score change)

SECONDARY OUTCOMES:
Change in Montgomery-Asberg Depression Rating Scale | week 0 (baseline), week 2, week 4 and week 6 (endpoint)
  Continuous measure (score changes)

CONTACTS AND LOCATIONS:
Overall Officials: Andre R Brunoni, MD, PhD, Principal Investigator — University of Sao Paulo
Locations (1):
- University Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Goerigk S, Cretaz E, Sampaio-Junior B, Vieira ELM, Gattaz W, Klein I, Lafer B, Teixeira AL, Carvalho AF, Lotufo PA, Bensenor IM, Buhner M, Padberg F, Brunoni AR. Effects of tDCS on neuroplasticity and inflammatory biomarkers in bipolar depression: Results from a sham-controlled study. Prog Neuropsychopharmacol Biol Psychiatry. 2021 Mar 8;105:110119. doi: 10.1016/j.pnpbp.2020.110119. Epub 2020 Oct 4. PMID 33022345
- [Derived] Tortella G, Sampaio-Junior B, Moreno ML, Moffa AH, da Silva AF, Lafer B, Lotufo PA, Gattaz W, Borrione L, Machado-Vieira R, Goerigk S, Bensenor IM, Brunoni AR. Cognitive outcomes of the bipolar depression electrical treatment trial (BETTER): a randomized, double-blind, sham-controlled study. Eur Arch Psychiatry Clin Neurosci. 2021 Feb;271(1):93-100. doi: 10.1007/s00406-020-01121-2. Epub 2020 Mar 27. PMID 32221654
- [Derived] Sampaio-Junior B, Tortella G, Borrione L, Moffa AH, Machado-Vieira R, Cretaz E, Fernandes da Silva A, Fraguas R, Aparicio LV, Klein I, Lafer B, Goerigk S, Bensenor IM, Lotufo PA, Gattaz WF, Brunoni AR. Efficacy and Safety of Transcranial Direct Current Stimulation as an Add-on Treatment for Bipolar Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):158-166. doi: 10.1001/jamapsychiatry.2017.4040. PMID 29282470
- See also: Website of Interdisciplinary Neuromodulation Service — http://www.sin.org.br